CLINICAL TRIAL: NCT02814942
Title: Prospective Evaluation of Asians With CRT for Heart Failure
Acronym: PEACH
Status: Recruiting | Type: Observational
Sponsor: National University Heart Centre, Singapore (Other)
Responsible Party: Principal Investigator, Pipin Kojodjojo, Consultant Cardiac Electrophysiologist, National University Heart Centre, Singapore
Other Study IDs: 2016/00608
Record Dates: First submitted 2016-06-22; First posted 2016-06-28 (Estimated); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Heart Failure; Cardiac Resynchronisation Therapy
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Years
Biospecimen Retention: Samples Without DNA — Serum saved for biomarking
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Heart Failure receiving CRT: Heart failure patients with QRS > 120ms receiving CRT
  Interventions: Device: Cardiac Resynchronization Therapy

INTERVENTIONS:
Device: Cardiac Resynchronization Therapy — Cardiac resynchronization therapy with or without ICD

SUMMARY:
Aim:To determine the baseline characteristics of heart failure patients in Singapore undergoing cardiac resynchronization therapy (CRT); the long term outcome and predictors of response to CRT.

Methodology:Among patients undergoing CRT for severe heart failure according to indications stipulated in international Cardiology guidelines, baseline demographic data is collected. Age, gender, NYHA functional class, co-morbidities, QRS width on ECG, presence of left bundle branch block pattern on ECG, presence of atrial fibrillation, left ventricular ejection fraction (LVEF) on echocardiogram, ventricular dimensions, 6 min walk test distance are collected. In addition, during the CRT implant procedure, blood is drawn from the vascular access and analysed for NT-pro BNP levels and other biomarkers of heart failure.

The echocardiographic and ECG parameters and blood biomarkers are reanalysed at 6 months and 12 months following CRT implant. Response to CRT is defined as a reduction in the iLVESV (left ventricular end-systolic volume index to body surface area) of >/= 15% and/or an increase in the LVEF of >/= 10%.

DETAILED DESCRIPTION:
Among patients undergoing CRT for severe heart failure according to indications stipulated in international Cardiology guidelines, baseline demographic data is collected. Age, gender, NYHA functional class, comorbidities, QRS width on ECG, presence of left bundle branch block pattern on ECG, presence of atrial fibrillation, left ventricular ejection fraction (LVEF) on echocardiogram, ventricular dimensions, 6 min walk test distance are collected. In addition, during the CRT implant procedure, blood is drawn from the vascular access and analysed for NT-pro BNP levels and other biomarkers of heart failure. The echocardiographic and ECG parameters and blood biomarkers are reanalysed at 6 months and 12 months following CRT implant. Response to CRT is defined as a reduction in the iLVESV (left ventricular end-systolic volume index to body surface area) of >/= 15% and/or an increase in the LVEF of >/= 10%.

ELIGIBILITY:
Inclusion Criteria:

* Broad QRS (>120 ms)
* EF < 40%
* Symptomatic heart failure
* Not on optimal medical therapy

Exclusion Criteria:

* Pregnant
* < 18 years of age
* Infection
* Unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Singaporean patients with broad QRS complexes, EF <40%, heart failure, requiring CRT
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2011-01; Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Echocardiographic response to CRT | 6 months
  A subject is considered an echocardiographic responder to CRT if there is:
  1. reduction in the iLVESV (left ventricular end-systolic volume index to body surface area) of >/= 15% OR
  2. an increase in the LVEF of >/= 10% during follow-up echocardiography at 6 months

SECONDARY OUTCOMES:
Neuroendocrine response to CRT | 6 months
  A subject is considered to have a neuro-endocrine response to CRT if BNP levels at 6 months post CRT implant has fallen more than 30% from baseline
Clinical response to CRT | 6 months
  A subject is considered a positive clinical responder to CRT if:
  1. NYHA class has improved by at least 1 class OR
  2. 6 minutes walking test has increased by at least 10%
Hospitalization For Cardiovascular events | 8 years
  Hospitalisation for acute coronary syndrome, heart failure, arrhythmias, ICD shocks or any unplanned admissions for any cardiac interventions or surgery
Mortality | 8 years
  Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Swee Chong Seow, MD, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No